CLINICAL TRIAL: NCT02305706
Title: Does Right Rather Than Left Starting Position Lead to Quicker Completion of COLonoscopy?
Brief Title: Right or Left for Colonoscopy?
Acronym: ROLCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ROLCOL 1.0
Record Dates: First submitted 2014-11-28; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Colonoscopy
Keywords: insertion; patient comfort
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right (Experimental): patients will be positioned on the right-lateral position at the start of colonoscopy
  Interventions: Procedure: starting position in colonoscopy
- Left (Active Comparator): patients will be positioned on the left-lateral position at the start of colonoscopy
  Interventions: Procedure: starting position in colonoscopy

INTERVENTIONS:
Procedure: starting position in colonoscopy

SUMMARY:
Colonoscopy is technically challenging. Conventionally, colonoscopy begins with patients positioned in the left lateral position. However, few published studies have explored alternatives and there is consequently little evidence to support left lateral starting position over alternatives.

DETAILED DESCRIPTION:
We aim to perform a randomised controlled trial of right versus left lateral starting position for colonoscopy. Primary outcome: time to caecum. Secondary outcomes: patient comfort; volume of sedation used.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age,
* informed consent,
* routine or urgent procedures

Exclusion Criteria:

* emergency colonoscopy,
* scheduled intubation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
time to caecum (insertion time from rectum to caecum) | 30 minutes
  insertion time from rectum to caecum

SECONDARY OUTCOMES:
patient comfort (visual analogue score) | 5 minutes
  patient comfort by visual analogue score

REFERENCES:
- [Derived] Vergis N, Scarborough AJ, Morris JA, Hoare JM. Prone or Left for Colonoscopy? A Randomized Controlled Trial of Prone Versus Left-sided Starting Position for Colonoscopy. J Clin Gastroenterol. 2018 Nov/Dec;52(10):e82-e86. doi: 10.1097/MCG.0000000000000871. PMID 28644314